CLINICAL TRIAL: NCT00280865
Title: Dose-Finding, Efficacy, and Safety of AZ 242 (Tesaglitazar) in Subjects With Type 2 Diabetes
Brief Title: GLAD: Dose-Finding, Efficacy, and Safety of AZ 242 (Tesaglitazar) in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-SBD-0001; GLAD
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2006-07-31 (Estimated); Status verified 2006-07

CONDITIONS: Type 2 Diabetes
Keywords: Tesaglitazar; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar; Pioglitazone; Diet

INTERVENTIONS:
Drug: Tesaglitazar
Drug: Pioglitazone
Behavioral: Dietary and Lifestyle Modification Counseling

SUMMARY:
This is a 12-week randomized, double-blind, multi-center, active-controlled (open-label pioglitazone) and placebo-controlled study of tesaglitazar (0.1, 0.5, 1, 2, and 3 mg) in patients with type 2 diabetes, not adequately controlled on diet and lifestyle advice alone during the run-in period. The study comprises a 2-week enrollment period, 4 week placebo single blind run in period followed by a 12-week double blind treatment period and a 3-week follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are 30 to 80 years of age
* Female patients: postmenopausal or surgically sterile
* Diagnosed with type 2 diabetes with C-peptide levels > 0.8 ng/mL
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), or to other PPAR g or PPAR a and g agonists.
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above 1.2 mg/dL
* Received any investigational product in other clinical studies within 30 days
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500
Dates: Start 2002-04; Study Completion 2003-06

PRIMARY OUTCOMES:
Absolute change from baseline to end of randomized treatment period in fasting plasma glucose (FPG)

SECONDARY OUTCOMES:
Changes in the following variables from baseline to the end of the randomized treatment period:
The change in plasma glucose and insulin during an oral glucose tolerance test
Insulin sensitivity by assessment of change in the calculated variable homeostasis assessment model
Lipid parameters (triglyceride [TG], total cholesterol, high-density lipoprotein cholesterol [HDL C], non-HDL C, low-density lipoprotein cholesterol [LDL C], apolipoproteins [Apo] A-I, Apo B, Apo CIII, free fatty acids
Change in insulin levels and hemoglobin A1c (HbA1c) levels
Responder analyses for FPG, TG, and HDL C according to pre-specified values
Pharmacokinetics of tesaglitazar
To assess the burden of type 2 diabetes mellitus in patients through the administration of the SF-36 health survey and the Well-Being Questionnaire (W BQ12) and comparing the study population data to published national and international normative data
To evaluate diabetes-specific instruments, Audit of Diabetes Dependent Quality of Life (ADDQoL) and The Diabetes Treatment Satisfaction Questionnaire (DTSQ) (s and c) in the study population and estimate the effect size of the instruments in patients r

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (110):
- United States (90):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Montgomery, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Alhambra, California
  - Research Site, Anaheim, California
  - Research Site, Dinuba, California
  - Research Site, Escondido, California
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, Long Beach, California
  - Research Site, Mission Viejo, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Walnut Creek, California
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Brandon, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, DeLand, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Blue Ridge, Georgia
  - Research Site, Dunwoody, Georgia
  - Research Site, Gurnee, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Bangor, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Salisbury, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Cadillac, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Henderson, Nevada
  - Research Site, Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canfield, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Lakewood, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Altoona, Pennsylvania
  - Research Site, Cheswick, Pennsylvania
  - Research Site, Penndel, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Warminster, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Columbia, South Carolina
  - Research Site, Ninety Six, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Arlington, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Lubbock, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Falls Church, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Edmonds, Washington
  - Research Site, Renton, Washington
  - Research Site, Huntington, West Virginia
- Canada (10):
  - Research Site, Edmonton, Alberta
  - Research Site, Burlington, Ontario
  - Research Site, Courtice, Ontario
  - Research Site, Granby, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Longueuil
  - Research Site, Montreal
  - Research Site, Sherbrooke
  - Research Site, Windsor
  - Research Site, Winnipeg
- France (7):
  - Research Site, Andard
  - Research Site, Angers
  - Research Site, Avrillé
  - Research Site, Chalonnes-sur-Loire
  - Research Site, Montrevault
  - Research Site, Segré
  - Research Site, Tiercé
- Mexico (3):
  - Research Site, Colonia del Valle
  - Research Site, Colonia Seccion XVI
  - Research Site, Delegacion Cuauhtemoc

REFERENCES:
- [Derived] Goldstein BJ, Rosenstock J, Anzalone D, Tou C, Ohman KP. Effect of tesaglitazar, a dual PPAR alpha/gamma agonist, on glucose and lipid abnormalities in patients with type 2 diabetes: a 12-week dose-ranging trial. Curr Med Res Opin. 2006 Dec;22(12):2575-90. doi: 10.1185/030079906x154169. PMID 17166340